CLINICAL TRIAL: NCT02414919
Title: Real-world Duration of Use for Highly Effective Reversible Contraception (HERC): A Retrospective Review
Brief Title: Duration of Use of Highly Effective Reversible Contraception
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: 17714
Record Dates: First submitted 2015-04-08; First posted 2015-04-13 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Pregnancy
MeSH Terms: interventions — Levonorgestrel; etonogestrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HERC: Women who had an insertion of HERC (Mirena IUD, ParaGard IUD, Implanon or Nexplanon)
  Interventions: Drug: Mirena (Levonorgestrel IUS, BAY86-5028); Drug: ParaGard; Drug: Implanon/Nexplanon

INTERVENTIONS:
Drug: Mirena (Levonorgestrel IUS, BAY86-5028) — Levonorgestrel-releasing intrauterine device 20 mcg/day
Drug: ParaGard — Copper T380A
Drug: Implanon/Nexplanon — Etonorgestrel contraceptive implant

SUMMARY:
To assess the proportion of women who use HERC for ≥2 years of duration

ELIGIBILITY:
Inclusion Criteria:

-Women who had an IUD or contraceptive implant inserted and removed within the University of Utah from January 1, 2004 to October 31, 2012

Ages: 15 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Women who had an IUD or contraceptive implant inserted at the University of Utah healthcare system
Sampling Method: Non-Probability Sample
Enrollment: 13880 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2016-03-28 (Actual); Study Completion 2016-03-28 (Actual)

PRIMARY OUTCOMES:
Proportion of women who use HERC | 2 years post-HERC initiation

SECONDARY OUTCOMES:
Duration of real world use of three different HERC devices | 2 years post-HERC initiation

OTHER OUTCOMES:
Difference in patient characteristics of women who chose different HERC devices | 2 years post-HERC initiation
Proportion of HERC used for ≥3 years of duration | ≥3 years post-HERC initiation
Model the predictors of ≥3 years of duration | ≥3 years post-HERC initiation

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Salt Lake City, Utah, United States

REFERENCES:
- [Background] Sanders J, Turok D, Gawron L, Law A, Wen L, Lynen R. Continuation of Long-Acting Reversible Contraception at Two Years in a University Healthcare Setting: A Retrospective Review. JMCP 2016;22(4a):S126
- [Result] Sanders JN, Turok DK, Gawron LM, Law A, Wen L, Lynen R. Two-year continuation of intrauterine devices and contraceptive implants in a mixed-payer setting: a retrospective review. Am J Obstet Gynecol. 2017 Jun;216(6):590.e1-590.e8. doi: 10.1016/j.ajog.2017.02.003. Epub 2017 Feb 8. PMID 28188772
- [Result] Sanders J, Turok D, Gawron L, Law A, Wen L, Lynen R. Three-Year Continuation of Long-Acting Reversible Contraceptive methods in a Mixed-Payer Health Care Setting: A Retrospective Review. Contraception 2016;94:405-406.